CLINICAL TRIAL: NCT05631158
Title: In Vivo Serial Neuromelanin MRI to Assess Depigmentation Rates in the Substantia Nigra of Early Parkinson's Disease
Brief Title: Neuromelanin MRI: A Progression Marker in Early PD
Acronym: InsIghtPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 281685
Record Dates: First submitted 2022-11-18; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-03

CONDITIONS: Parkinson Disease; Progression, Disease
MeSH Terms: conditions — Parkinson Disease; Disease Progression | interventions — Hematologic Tests; Physical Examination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early Parkinson's disease: All the participants will undergo five clinical examination, four MRI scans and one fasting blood test in total in this serial study.
  Interventions: Diagnostic Test: MRI
- Healthy Controls: This cohort will undergo the same procedure of the patient's group.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — The clinical examination includes a short physical exam, a brief history of allergies, previous diseases and medications, and disease-related questionnaires.
  All the participants will undergo 4 serial MRI scans: one MRI scan at the baseline visit, 6, 12, 18 months follow-up visit, respectively to record the changes in the brain, which include the neuromelanin scan.
  For future proving the value of our study, we will also collect and store blood samples at the initial visit.
  Other Names: Blood test; Physical examination

SUMMARY:
Prospective observational study to qualify NM-MRI as progression marker in early Parkinson's.

DETAILED DESCRIPTION:
Parkinson's is the second most common neurodegenerative disorder with progressive, disabling motor and non- motor symptoms for which effective symptomatic, but non disease-modifying treatment is available. Neuromelanin- containing neurons in the substantia nigra undergo neurodegeneration during Parkinson's disease. There is considerable heterogeneity in the progression of cell loss and clinical symptoms with major research interest in identifying prognostic subtypes.

A non-invasive biomarker that can track the loss of the neuromelanin-containing neurons would be highly desirable to (i) study subtype-specific trajectories of SN depigmentation, (ii) track disease progression in early Parkinson's to assist in stratifying groups and outcome assessment in clinical intervention trials, and (iii) enable patients and their families to better manage their condition including informed forward planning. Neuromelanin MRI (NM-MRI) is a new approach sensitive to the neuromelanin-iron complex, with proven association with the tissue changes of the number of the neuromelanin-containing neurons. Its diagnostic value was established in several studies case-control, but there is a lack of standardisation, multi-centre studies and prospective diagnostic trials. To date only a small, single arm retrospective study reported serial NM loss in Parkinson's.

Building on our previous work, the proposed research entails the development of an early progression biomarker for Parkinson's disease that is pathologically relevant, non-invasive, and uses MRI which is a widely available imaging method for detection. The experimental approach combines advanced computational imaging, retrospective use and extension of existing cohorts with a new dedicated prospective serial study using NM-MRI in uncertain parkinsonism, de novo and early Parkinson and healthy controls using latest MRI technology.

ELIGIBILITY:
Inclusion Criteria:

-Inclusion criteria for patients:

* For Parkinson's patients and early-onset Parkinson's:

  1. Diagnosis of Parkinson's disease, based on UK Brain Bank criteria and made within the preceding 3 years ('recent onset cases'); or
  2. diagnosed at under 50 years ('under 50 years cases')
* For clinical symptoms suspicious for a diagnosis of PD but clinical uncertainty with regard to a definite diagnosis:

  1. clinical symptoms not meeting all of the required UK Brain Bank diagnostic criteria for the diagnosis of PD; or
  2. clinical features not typically associated with PD and therefore raising the possibility of a different type disorder/movement disorder referred for a DaTSCAN as part of the National Health Service (NHS) clinical diagnostic work-up to investigate a suspicion for a parkinsonian movement disorder-type disease, or referred for a research DaTSCAN as part of existing N3iPD and PaMIR studies for the diagnostic work-up to investigate a suspicion for a parkinsonian movement disorder-type disease.
* Age ≥18 to <90years
* Being able and willing to provide informed consent

Inclusion criteria for healthy controls:

* Age ≥18 to <90years
* Being able and willing to provide informed consent

Exclusion Criteria:

* Exclusion criteria for patients:

  1. The patient has severe comorbid illness that would prevent full study participation
  2. The patient has features indicating another type of degenerative parkinsonism, e.g. progressive supranuclear palsy
  3. Drug-induced parkinsonism (Drug-unmasked PD is allowed)
  4. Symmetrical lower body parkinsonism attributable to significant cortical and/or subcortical cerebrovascular disease (patients with 'incidental' small vessel disease on brain imaging are allowed).
  5. Negative or normal functional imaging of the presynaptic dopamine system
  6. The presence of UK Brain Bank exclusion criteria will be recorded at baseline, allowing for the presence of 1 or 2 exclusion criteria (e.g. dopamine antagonist Drug used; more than one affected relative) (if justified e.g. by abnormal SPECT).
  7. Any contraindication to Magnetic Resonance (MR) scanning.
  8. Any major neurological (other than PD), psychiatric or cardiovascular disease or history of brain injury.
  9. Medical illness or medication that may affect brain morphometry or function.
  10. Patient who is pregnant and/or breastfeeding.

Exclusion criteria for healthy controls:

1. Subject has severe comorbid illness that would prevent study participation
2. Subject already has a diagnosis of Parkinson's disease
3. Any contraindication to Magnetic Resonance (MR) scanning
4. Subject who is pregnant and/or breastfeeding.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All potential participants need to have to capacity to give consent prior to study enrolment. Study participation is not possible if the participant is unable to give consent or does not have the capacity to consent.
Sampling Method: Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Neuromelanin signal in PD | 6 months
  The primary outcome measure of this study is the neuromelanin-related signal on dedicated 3T MRI.

SECONDARY OUTCOMES:
Depigmentation rates | 2 years
  * differences in depigmentation rates between Parkinson's and controls in extended retrospective cohorts (discovery)
  * to assess whether earlier depigmentation rates can predict longer term clinical change based on commonly used outcome markers in clinical trials

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
A new high-quality neuromelanin MRI database with linked whole brain multimodal MRI, clinical findings and stored blood samples. We intend to quality control and curate the imaging and clinical data for the generation of a data repository, and have included cost for data storage, but ultimately intend to integrate this into the Critical Pathway Initiative. Where possible. We also aim to release imaging-derived parameters to make the data usable for non-imaging communities.
Supporting Information: Analytic Code
Time Frame: within 5 years
Access Criteria: Open access